CLINICAL TRIAL: NCT02193828
Title: A Phase 2a, Double-blind, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Effectiveness of AA4500 in the Treatment of Dupuytren's Disease Nodules
Brief Title: Phase 2a Dose-Ranging Study to Evaluate Safety and Effectiveness of AA4500 in Treatment of Dupuytren's Disease Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUX-CC-750
Record Dates: First submitted 2014-06-19; First posted 2014-07-18 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Dupuytren's Disease
Keywords: Dupuytren's nodules
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AA4500 0.25 mg (Experimental): Collagenase clostridium histolyticum, single 0.25 mg injection
  Interventions: Biological: Collagenase clostridium histolyticum
- AA4500 0.40 mg (Experimental): Collagenase clostridium histolyticum, single 0.40 mg injection
  Interventions: Biological: Collagenase clostridium histolyticum
- AA4500 0.60 mg (Experimental): Collagenase clostridium histolyticum, single 0.60 mg injection
  Interventions: Biological: Collagenase clostridium histolyticum
- Placebo (Placebo Comparator): Placebo, single 0.25 mg, 0.40 mg, or 0.60 mg injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Collagenase clostridium histolyticum — Single injection into nodule
  Other Names: AA4500; XIAFLEX; XIAPEX
  Arms: AA4500 0.25 mg; AA4500 0.40 mg; AA4500 0.60 mg
Biological: Placebo — Single injection into nodule
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the safety and effectiveness of AA4500 in treating palmar Dupuytren's disease nodules.

DETAILED DESCRIPTION:
Approximately 13 sites in the United States and Australia, approximately 90 study subjects.

After all pre-injection procedures are completed on day 1, eligible men and women will be randomized in a 1:1:1 ratio to dose group and then in a 4:1 ratio to treatment group. Study drug will be administered into a palmar nodule located on the selected hand.

AA4500 (collagenase clostridium histolyticum) 3 doses (low, medium, and high) after reconstitution with sterile diluent (0.3 mg/mL calcium chloride dihydrate in 0.9% sodium chloride). Each dose of study drug will be injected into the nodule. The injection will be administered in 3 different volumes according to randomization.

Placebo after reconstitution with sterile diluent (0.3 mg/mL calcium chloride dihydrate in 0.9% sodium chloride). Each dose of study drug will be injected into the nodule. The injection will be administered in 3 different volumes according to randomization.

Follow up visits for the evaluation of safety and efficacy will be required for all subjects on days 8, 29, and 57.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent
2. Be a man or woman ≥ 18 years of age
3. Have a diagnosis of Dupuytren's disease AND have at least one palmar nodule on the selected hand that is:

   1. Palpable
   2. Measures between 0.5 cm and 2.0 cm in length and between 0.5 cm and 2.0 cm in width using hand-held calipers n
   3. Not directly associated with a Dupuytren's cord
4. Have a negative urine pregnancy test at screening and before injection of study drug and be using a highly effective (ie, < 1% failure rate) contraception method as judged by the investigator (eg, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for the duration of the study or be surgically sterile (if female of childbearing potential); or be a postmenopausal female (no menses for at least 1 year or hysterectomy)
5. Be able to comply with the study visit schedule as specified in the protocol

Exclusion Criteria:

1. Received steroid injections (eg, tri-amcinolone acetonide) on the selected nodule within 3 months before administration of study drug
2. Has a chronic muscular, neurological, or neuromuscular disorder that affects the hands
3. Has a known systemic allergy to collagenase or any other excipient of AA4500
4. Has received any collagenase treatments (eg, Santyl® ointment and/or XIAFLEX®/XIAPEX®) within 30 days before injection of study drug in the hand selected for treatment
5. Is currently receiving or plans to receive anticoagulant medication or has received anticoagulant medication (except for ≤ 150 mg aspirin daily) within 7 days before injection of study drug
6. Has a known recent history of stroke, bleeding, or other medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
7. Received an investigational drug within 30 days before injection of study drug
8. Is pregnant or intends on becoming pregnant during the study or is breastfeeding a child
9. Has any clinically significant medical history or condition(s), including conditions that affect the hands, that would, in the opinion of the investigator, substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives of the study
10. Had surgery on the selected hand within 3 months before the screening visit
11. Has jewelry on the hand to be treated that cannot be removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD MPH, Study Director — Endo Pharmaceuticals
Locations (11):
- United States (9):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Brigid Freyne, MD, Inc., Murrieta, California
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - State University of New York, Stony Brook, New York
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Orthopedic and Reconstructive Center, Oklahoma City, Oklahoma
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
- Australia (2):
  - Brisbane Hand & Upper Limb Clinic, Brisbane, Queensland
  - Houston Medical, Kippa-Ring, Queensland

REFERENCES:
- [Derived] Costas B, Coleman S, Kaufman G, James R, Cohen B, Gaston RG. Efficacy and safety of collagenase clostridium histolyticum for Dupuytren disease nodules: a randomized controlled trial. BMC Musculoskelet Disord. 2017 Aug 30;18(1):374. doi: 10.1186/s12891-017-1713-z. PMID 28854973

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.60 mg: Collagenase clostridium histolyticum (AA4500), single 0.60 mg injection into the nodule
- AA4500 0.40 mg: Collagenase clostridium histolyticum (AA4500), single 0.40 mg injection into the nodule
- AA4500 0.25 mg: Collagenase clostridium histolyticum (AA4500), single 0.25 mg injection into the nodule
- Placebo: Placebo, single 0.25 mg, 0.40 mg, or 0.60 mg injection into the nodule
Period: Overall Study
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Started | 18 | 18 | 23 | 17
Completed | 18 | 18 | 22 | 16
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis based on Safety population; all randomized subjects who received an injection of study medication. One subject did not receive study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 22 | 17 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 16 | 11 | 52
  >=65 years | 5 | 6 | 6 | 6 | 23
Age, Continuous [Median (Full Range); unit: years] | 62.0 [41 to 84] | 60.0 [37 to 75] | 57.0 [32 to 73] | 58.0 [45 to 73] | 58.0 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 11 | 7 | 34
  Male | 12 | 8 | 11 | 10 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 17 | 17 | 21 | 16 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 18 | 17 | 22 | 17 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 14 | 12 | 48
  Australia | 6 | 8 | 8 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Surface Area and Volume of the Treated Nodule at Day 57 Using Caliper Measurements
Description: Percent change from baseline in surface area and volume of the treated nodule was determined from hand-held caliper measurements of the length and width of the nodule. Percent change = 100*(Day 57 area [or volume] - baseline area [or volume])/baseline area [or volume]. A negative value represents the improvement from baseline (decreased size) while a positive value represents worsening.
Time Frame: Baseline, Day 57
Population: Analysis based on Modified Intent-to-Treat (mITT) population; all randomized subjects who received study medication and had pre- and post-baseline nodule measurements for ultrasound and calipers. Analytical outliers (subjects whose percent change in ultrasound volume was greater than the 75th percentile + 3× the interquartile range) were excluded.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 17 | 18 | 20 | 15
percentage of change
  Surface Area | -81.61 (20.251) | -80.11 (21.459) | -58.30 (29.849) | -41.76 (32.445)
  Volume | -89.03 (15.016) | -87.58 (16.372) | -68.15 (33.859) | -49.13 (36.736)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; For surface area; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; For surface area; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; For surface area; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; For surface area; Test type: Superiority or Other; p = .0713, ANOVA
Statistical Analysis 5: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; For volume; Test type: Superiority or Other; p = .0002, ANOVA
Statistical Analysis 6: Comparison: AA4500 0.60 mg vs Placebo; For volume; Test type: Superiority or Other; p = .0001, ANOVA
Statistical Analysis 7: Comparison: AA4500 0.40 mg vs Placebo; For volume; Test type: Superiority or Other; p = .0001, ANOVA
Statistical Analysis 8: Comparison: AA4500 0.25 mg vs Placebo; For volume; Test type: Superiority or Other; p = .0446, ANOVA

2. Secondary Outcome: Percent Change From Baseline in Surface Area and Volume of the Treated Nodule at Day 57 Using Ultrasound
Description: Percent change from baseline in surface area and volume of the treated nodule was determined from ultrasound measurements of the length, width, and depth of the nodule. Percent change = 100*(Day 57 area [or volume] - baseline area [or volume])/baseline area [or volume]. A negative value represents the improvement from baseline (decreased size) while a positive value represents worsening.
Time Frame: Baseline, Day 57
Population: Analysis based on mITT population; all randomized subjects who received study medication and had pre- and post-baseline nodule measurements for ultrasound and calipers. Analytical outliers (subjects whose percent change in ultrasound volume was greater than the 75th percentile + 3× the interquartile range) were excluded.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 17 | 18 | 20 | 15
percentage of change
  Surface Area | -34.23 (41.353) | -19.37 (39.658) | -10.30 (41.696) | -4.54 (54.784)
  Volume | -40.99 (46.612) | -13.01 (68.804) | -9.52 (60.156) | -7.19 (69.877)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; For surface area; Test type: Superiority or Other; p = .2431, ANOVA
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; For surface area; Test type: Superiority or Other; p = .0625, ANOVA
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; For surface area; Test type: Superiority or Other; p = .3409, ANOVA
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; For surface area; Test type: Superiority or Other; p = .7040, ANOVA
Statistical Analysis 5: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; For volume; Test type: Superiority or Other; p = 0.3556, ANOVA
Statistical Analysis 6: Comparison: AA4500 0.60 mg vs Placebo; For volume; Test type: Superiority or Other; p = .1275, ANOVA
Statistical Analysis 7: Comparison: AA4500 0.40 mg vs Placebo; For volume; Test type: Superiority or Other; p = .7883, ANOVA
Statistical Analysis 8: Comparison: AA4500 0.25 mg vs Placebo; For volume; Test type: Superiority or Other; p = .9123, ANOVA

3. Secondary Outcome: Change From Baseline in Consistency of the Treated Nodules at Day 57
Description: Investigators determined the consistency of the nodule through palpitation using a 5-point scale: 5 = hard (solid), 4 = firm throughout, 3 = moderate firmness, 2 = soft, and 1 = non-palpable. The change scores could range from +4 (greatest worsening in consistency) to -4 (greatest improvement in consistency); a negative change from baseline value reflects improvement from baseline (softening) while a positive value reflects worsening.
Time Frame: Baseline, Day 57
Population: Analysis based on mITT population; all randomized subjects who received an injection of study medication and had pre- and post-baseline nodule measurements for both ultrasound and calipers. Subjects with an incomplete assessment (not done) on Day 57 were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 16 | 17 | 22 | 15
units on a scale | -1.9 (0.93) | -1.9 (1.05) | -1.2 (1.10) | -0.3 (0.96)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0002, Kruskal-Wallis
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p < .0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p = .0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0139, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percent Change From Baseline in Hardness of the Treated Nodule at Day 57
Description: A durometer was used to assess nodule hardness on a scale of 0 (soft) to 100 (hard). Percent change = 100*(Day 57 hardness - baseline hardness)/baseline hardness. A negative value represents the improvement from baseline (softening) while a positive value represents worsening.
Time Frame: Baseline, Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 16 | 17 | 22 | 15
percentage of change | -17.05 (15.584) | -30.40 (24.930) | -17.87 (22.265) | 4.80 (23.959)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0004, ANOVA
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p = .0075, ANOVA
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0031, ANOVA

5. Secondary Outcome: Change From Baseline in Nodular Pain of the Treated Nodule at Day 57
Description: After the nodule was squeezed using a dynamometer, subjects were asked to rate the amount of pain they felt on an 11-point visual analog scale (VAS) from 0 (no pain or discomfort) to 10 (extreme pain or discomfort). A negative change from baseline value reflects improvement from baseline (less pain) while a positive value reflects worsening.
Time Frame: Baseline, Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 16 | 17 | 22 | 15
units on a scale | -0.8 (1.97) | -1.6 (2.21) | -1.7 (2.57) | -0.5 (1.77)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .3135, ANOVA
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p = .7249, ANOVA
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p = .1573, ANOVA
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .1234, ANOVA

6. Secondary Outcome: Investigator Global Assessment of Improvement With Treatment
Description: Investigators were asked to determine the degree of improvement in the subject's treated nodule compared with screening on a 7-point scale: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Day 57
Population: Analysis based on mITT population; all randomized subjects who received an injection of study medication and had pre- and post-baseline nodule measurements for both ultrasound and calipers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 22 | 16
units on a scale | 1.7 (0.84) | 1.7 (0.75) | 2.5 (1.10) | 3.0 (1.15)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0006, Kruskal-Wallis
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p = .0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p = .0012, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .1298, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Subject Satisfaction With Treatment
Description: Subjects were asked to rate their satisfaction with treatment on a 5-point scale: 1 = very satisfied, 2 = quite satisfied, 3 = neither satisfied nor dissatisfied, 4 = quite dissatisfied, and 5 = very dissatisfied.
Time Frame: Day 57
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 22 | 16
units on a scale | 1.5 (0.79) | 1.6 (0.85) | 2.3 (1.17) | 2.8 (1.34)
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0048, Kruskal-Wallis
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p = .0034, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p = .0079, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .3216, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Composite Responder Analysis
Description: A composite responder is a subject who had an improved assessment [values of 1 (very much improved), 2 (much improved), or 3 (minimally improved)] on the investigator global assessment and had a satisfied assessment [values of 1 (very satisfied) or 2 (quite satisfied)] on the subject assessment.
Time Frame: Day 57
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 22 | 16
participants
  Responder: Yes | 14 | 16 | 12 | 6
  Responder: No | 4 | 2 | 10 | 10
Statistical Analysis 1: Comparison: AA4500 0.60 mg vs AA4500 0.40 mg vs AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .0065, Fisher Exact
Statistical Analysis 2: Comparison: AA4500 0.60 mg vs Placebo; Test type: Superiority or Other; p = .0349, Fisher Exact
Statistical Analysis 3: Comparison: AA4500 0.40 mg vs Placebo; Test type: Superiority or Other; p = .0033, Fisher Exact
Statistical Analysis 4: Comparison: AA4500 0.25 mg vs Placebo; Test type: Superiority or Other; p = .3423, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through the end of the study (Day 57).
Description: Adverse events are reported for the Safety population; all randomized subjects who received an injection of study medication.
Arm/Group | AA4500 0.60 mg | AA4500 0.40 mg | AA4500 0.25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/22 | 0/17
Other Adverse Events (participants affected / at risk) | 17/18 | 18/18 | 21/22 | 7/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AA4500 0.60 mg (N=18) | AA4500 0.40 mg (N=18) | AA4500 0.25 mg (N=22) | Placebo (N=17)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 4 | 1 | 6 | 0
Injection site bruising (General disorders) | 6 | 4 | 5 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 2 | 0
Injection site hypoaesthesia (General disorders) | 1 | 0 | 0 | 0
Injection site oedema (General disorders) | 2 | 0 | 2 | 0
Injection site pain (General disorders) | 2 | 4 | 4 | 0
Injection site pruritus (General disorders) | 2 | 3 | 2 | 1
Injection site swelling (General disorders) | 0 | 4 | 5 | 0
Local swelling (General disorders) | 10 | 7 | 8 | 3
Localised oedema (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Tenderness (General disorders) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 9 | 9 | 13 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 10 | 10 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other